CLINICAL TRIAL: NCT00594815
Title: A Pilot Study of Combined Immunochemotherapy Followed by Reduced Dose RT for Patients With Newly Diagnosed Primary Central Nervous System Lymphoma
Brief Title: Combined Immunochemotherapy Followed By Reduced Dose Radiation Therapy (RT) for Patients With Newly Diagnosed Primary Central Nervous System Lymphoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Northwestern Memorial Hospital (Other); Columbia University (Other); Kentuckiana Cancer Institute (Other); University of Virginia (Other); University of Vermont (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 01-146; NCT00059956 (obsolete NCT alias)
Record Dates: First submitted 2008-01-07; First posted 2008-01-16 (Estimated); Results first posted 2017-04-06 (Actual); Last update posted 2017-04-06 (Actual); Status verified 2017-04

CONDITIONS: Lymphoma
Keywords: Lymphoma; Central Nervous System
MeSH Terms: conditions — Lymphoma | interventions — Cytarabine; Leucovorin; Methotrexate; Procarbazine; Rituximab; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Cytarabine, Leucovorin, Methotrexate, Procarbazine, Rituximab, Vincristine

INTERVENTIONS:
Drug: Cytarabine, Leucovorin, Methotrexate, Procarbazine, Rituximab, Vincristine — Immunochemotherapy

SUMMARY:
The purpose of this study is to find out if immunotherapy (rituximab) added to chemotherapy is a safe treatment for primary central nervous system lymphoma (PCNSL). PCNSL is a rare tumor. It is usually treated with chemotherapy and radiation. This combination prolongs survival, but about half of patients relapse. The investigators hope that the addition of rituximab will improve the control of the tumor.

DETAILED DESCRIPTION:
The purpose of this study is to find out if immunotherapy (rituximab) added to chemotherapy is a safe treatment for primary central nervous system lymphoma (PCNSL). PCNSL is a rare tumor. It is usually treated with chemotherapy and radiation. This combination prolongs survival, but about half of patients relapse. We hope that the addition of rituximab will improve the control of your tumor.

The second goal of this study is to assess a lower dose of brain radiation. Brain radiation may cause memory loss or dementia. For patients over the age of 60, the risk of significant memory loss is 80-90%. The risk for younger patients is smaller but less clear. In this, study patients whose tumors are in remission after chemotherapy will be treated with a lower dose of brain radiation. We hope that this lower dose will be less toxic. However, it is also possible that using a lower dose of radiation will be less effective in controlling your tumor.

ELIGIBILITY:
Inclusion Criteria:

* All patients must have a histologic diagnosis of non-Hodgkin's lymphoma by brain biopsy. Patients who have an inconclusive biopsy or who are not candidates for biopsy may be eligible provided they have a typical cranial magnetic resonance imaging (MRI) or computed tomography (CT) scan and meet at least one of the following two criteria:

  * A positive cerebrospinal fluid (CSF) cytology for lymphoma or a monoclonal lymphocyte population as defined by cell surface markers
  * A biopsy of the vitreous or uvea demonstrating non-Hodgkin's lymphoma
* A typical MRI/CT scan for primary intracranial lymphoma is defined as the presence of hypo, iso, or hyperdense parenchymal contrast-enhancing (usually homogeneously) mass lesion(s)
* Patients must be HIV-1 negative
* Patients must have a normal or negative pre-treatment systemic evaluation including:

  * A bone marrow aspirate and biopsy
  * CT scans of the chest, abdomen and pelvis
  * Patients must have adequate bone marrow function (defined as peripheral leucocyte count > 4000 cells/mm3 and platelet count > 100,000 cells/mm3), liver function (bilirubin < 2.0 mg and SGOT < 2 times upper limit of normal), and adequate renal function (serum creatinine < 1.5 mg/dl or creatinine clearance > 50 cc/min/1.73M2)
* Men and women of reproductive potential must agree to use an acceptable method of birth control during treatment and for six months after completion of treatment

Exclusion Criteria:

The following would exclude a patient from the study:

* Prior cranial irradiation
* Other active primary malignancy with the exception of basal cell carcinoma of the skin and cervical carcinoma in situ
* Pre-existing immunodeficiency such as renal transplant recipient
* Prior treatment with chemotherapy for CNS lymphoma

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2002-08-28; Primary Completion 2016-02-23 (Actual); Study Completion 2016-02-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Omuro, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] Morris PG, Correa DD, Yahalom J, Raizer JJ, Schiff D, Grant B, Grimm S, Lai RK, Reiner AS, Panageas K, Karimi S, Curry R, Shah G, Abrey LE, DeAngelis LM, Omuro A. Rituximab, methotrexate, procarbazine, and vincristine followed by consolidation reduced-dose whole-brain radiotherapy and cytarabine in newly diagnosed primary CNS lymphoma: final results and long-term outcome. J Clin Oncol. 2013 Nov 1;31(31):3971-9. doi: 10.1200/JCO.2013.50.4910. Epub 2013 Oct 7. PMID 24101038
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Protocol Open to Accrual 08/08/2002 Protocol Closed to Accrual 03/10/2009 Primary Completion Date 02-23-2016 Recruitment Location is the medical clinic
Groups:
- Immunocompetent Pts With Newly Diagnosed Primary CNS Lymphoma: Cytarabine, Leucovorin, Methotrexate, Procarbazine, Rituximab, Vincristine: Immunochemotherapy
Period: Overall Study
Arm/Group | Immunocompetent Pts With Newly Diagnosed Primary CNS Lymphoma
Started | 52
Completed | 43
Not Completed | 9
Not completed — Never Treated | 3
Not completed — Withdrawal by Subject | 2
Not completed — Toxicity | 4

BASELINE CHARACTERISTICS:
Arm/Group | Immunocompetent Pts With Newly Diagnosed Primary CNS Lymphoma
Number analyzed (Participants) | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 34
  >=65 years | 18
Age, Continuous [Median (Full Range); unit: Years] | 60 [30 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 30

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Participants Who Experienced Acute Treatment Related Adverse Events
Description: The toxicity of this combined regimen will be measured using the NCI CTC version 2.0.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Immunocompetent Pts With Newly Diagnosed Primary CNS Lymphoma
Number analyzed (Participants) | 52
Participants | 52

2. Primary Outcome: Progression Free Survival
Description: Overall Progression Free Survival at 2 years
Time Frame: 2 Years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Immunocompetent Pts With Newly Diagnosed Primary CNS Lymphoma
Number analyzed (Participants) | 52
percentage of participants | 57 [44 to 71]

ADVERSE EVENTS:
Time Frame: Every other week during treatment cycles. Follow up evaluation will be assessed every 3 months for the first year after completing treatment. Follow up will then be done every 4 months for the second year, every 6 months until the 5th year and then annually.
Groups:
- Immunocompetent Pts With Newly Diagnosed Primary CNS Lymphoma: This is a single-armed pilot study designed to evaluate the safety and efficacy of combined immunochemotherapy followed by reduced dose radiation for participants with newly diagnosed PCNSL.
Arm/Group | Immunocompetent Pts With Newly Diagnosed Primary CNS Lymphoma
All-Cause Mortality (participants affected / at risk) | 13/52
Serious Adverse Events (participants affected / at risk) | 22/52
Other Adverse Events (participants affected / at risk) | 43/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Immunocompetent Pts With Newly Diagnosed Primary CNS Lymphoma (N=52)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Ataxia (Nervous system disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Elevated Creatinine (Renal and urinary disorders) | 1
Dehydration (Gastrointestinal disorders) | 1
Duodenal ulcer (Gastrointestinal disorders) | 1
Febrile neutropenia (Infections and infestations) | 3
Fever (General disorders) | 2
Hallucinations (Psychiatric disorders) | 1
Hypotension (Cardiac disorders) | 2
Infection without neutropenia (Infections and infestations) | 4
Infection (Infections and infestations) | 1
Leukocytes (Blood and lymphatic system disorders) | 4
Mood alteration-anxiety (Psychiatric disorders) | 1
Mood alteration - depression (Psychiatric disorders) | 1
Radiation mucositis (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Neurology, other (Nervous system disorders) | 2
Neutrophils/granulocytes (Investigations) | 4
Pain, other (General disorders) | 1
Personality/behavior (Psychiatric disorders) | 1
Platelets (Investigations) | 4
Pulmonary, other (Respiratory, thoracic and mediastinal disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Renal/GU, other (Renal and urinary disorders) | 1
Thrombosis (Vascular disorders) | 1
Vision-double vision (Eye disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Wound, infectious (Infections and infestations) | 3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Immunocompetent Pts With Newly Diagnosed Primary CNS Lymphoma (N=52)
Hypocalcemia (Metabolism and nutrition disorders) | 36
Hyperglycemia (Metabolism and nutrition disorders) | 36
Hemoglobin/Anemia (Blood and lymphatic system disorders) | 33
Leukocytes (Immune system disorders) | 31
SGPT (ALT) (Investigations) | 24
Lymphopenia (Immune system disorders) | 30
Neutrophils/granulocytes (Investigations) | 22
SGOT (AST) (Investigations) | 16
Platelets (Investigations) | 14
Hypophosphatemia (Metabolism and nutrition disorders) | 10
PT (Investigations) | 9
Hypoalbuminemia (Metabolism and nutrition disorders) | 8
Hyponatremia (Metabolism and nutrition disorders) | 7
Hypokalemia (Metabolism and nutrition disorders) | 7
PTT (Investigations) | 6
Creatinine (Renal and urinary disorders) | 6
Constipation (Gastrointestinal disorders) | 5
Bilirubin (Hepatobiliary disorders) | 5
Hypoglycemia (Metabolism and nutrition disorders) | 4
Fatigue (General disorders) | 4
Hyperkalemia (Metabolism and nutrition disorders) | 3
Neuropathy-sensory (Nervous system disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes